CLINICAL TRIAL: NCT03256045
Title: CLBH589DUS108T: Panobinostat With Carfilzomib and Dexamethasone for Relapsed/Refractory Multiple Myeloma: Correlation With In Vitro Chemosensitivity Testing
Brief Title: Panobinostat, Carfilzomib, and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to loss of funding and former PI left the institution
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH); SecuraBio (Industry)
Responsible Party: Principal Investigator, Andrew Cowan, Assistant Professor, Division of Medical Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9757; NCI-2017-00453 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9757 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1016013 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment-panobinostat, carfilzomib, dexamethasone,chemo assay (Experimental): Patients receive panobinostat PO on days 1, 3, 5, 15, 17, and 19. Patients also receive carfilzomib IV and dexamethasone PO on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and/or bone marrow samples for testing via in vitro chemosensitivity assay.
  Interventions: Drug: Carfilzomib; Other: Chemosensitivity Assay; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Panobinostat

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Other: Chemosensitivity Assay — Undergo in vitro chemosensitivity testing
  Other Names: Chemosensitivity Testing
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Panobinostat — Given PO
  Other Names: Faridak; Farydak; LBH589

SUMMARY:
This phase II trial studies how well panobinostat, carfilzomib, and dexamethasone work in treating patients with multiple myeloma that has come back (relapsed) or does not respond to treatment (refractory). Panobinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as carfilzomib and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Using multiple myeloma cells from patients' blood samples, the researchers will do laboratory tests to look at how well each of the drugs, alone and in different combinations, kill multiple myeloma cells. If the laboratory tests work well, they may be used in the future to help plan treatment for future patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To correlate in vitro drug sensitivity testing with clinical response by determining the rate of in vitro drug sensitivity to panobinostat, carfilzomib, and dexamethasone singly and in combination, doublets and triplets.

SECONDARY OBJECTIVE:

I. To monitor response rates (partial response [PR], very good partial response [VGPR], and complete response) using the International Myeloma Working Group Uniform Response Criteria for Multiple Myeloma.

EXPLORATORY OBJECTIVE:

I. Progression free survival and overall survival will be assessed for up to 3 years after last dose.

OUTLINE:

Patients receive panobinostat orally (PO) on days 1, 3, 5, 15, 17, and 19. Patients also receive carfilzomib intravenously (IV) and dexamethasone PO on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood and/or bone marrow samples for testing via in vitro chemosensitivity assay.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma refractory to or relapsed after >= 1 line of prior therapy (International Myeloma Working Group [IMWG] criteria)
* Measurable disease, as indicated by one of the following:

  * Serum monoclonal (M)-protein >= 1.0 g/dL
  * Elevated involved free light chain >= 10 mg/dL as per IMWG criteria, and abnormal ratio
  * Urine Bence Jones protein > 200 mg/24 hour (hr)
* Absolute neutrophil count (ANC) >= 750/uL
* Platelet count >= 75,000/uL
* Hemoglobin >= 7 g/dL
* Creatinine =< 2.0 mg/dL or calculated creatinine clearance >= 30 mL/min
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless elevation is thought to be due to Gilbert's syndrome
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SPGT) (alanine aminotransferase [ALT]) =< 2.5 x ULN
* Patients must avoid consumption of grapefruit, pomegranates, starfruit, Seville oranges or products containing the juice of each during the entire study and preferably 7 days before the first dose of study medications; orange juice is allowed
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, should have a pregnancy test prior to the initiation of treatment and use highly effective methods of contraception during and for 3 months post study treatment; highly effective contraception methods include total abstinence, female sterilization, male sterilization, use of oral, injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy; women using hormonal contraceptives should additionally use a barrier method of contraception; women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural amenorrhea or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks ago
* Sexually active males must use a condom during intercourse while taking study drug and for 6 months after stopping treatment; males should not father a child in this period; a condom is required to be used also by vasectomized men as well as during intercourse with a male partner; female partners of sexually active men should also use an effective contraception during treatment and for 6 months after their male partner has stopped taking the drug

Exclusion Criteria:

* Another bone marrow malignancy
* Another cancer with expected survival of < 2 years
* Active viral, bacterial, or fungal infection progressing on current treatment
* Clinically significant uncontrolled heart disease and/or recent cardiac event within 6 months prior to enrollment, such as:

  * History of angina pectoris, symptomatic pericarditis, or myocardial infarction
  * Left ventricular ejection fraction (LVEF) < 45% as determined by echocardiogram (ECHO) or multi gated acquisition (MUGA) scan
  * History or presence of any significant, uncontrolled, or persistent cardiac arrhythmias, e.g. ventricular, supraventricular, nodal arrhythmias or conduction abnormality; stable atrial fibrillation within 6 months prior to randomization is permitted
  * Presence of unstable atrial fibrillation (ventricular response rate > 100 beats per minute [bpm]); NOTE: patients with stable atrial fibrillation can be enrolled provided they do not meet other cardiac exclusion criteria
  * Resting heart rate < 50 bpm
  * Complete left bundle branch block (LBBB), bifascicular block
  * Congenital long QT syndrome
  * Any clinically significant ST segment and/or T-wave abnormalities
  * Corrected QT (QTcF) > 450 msec for males and > 470 msec for females using Fridericia's correction on screening electrocardiogram (ECG)
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Uncontrolled hypertension defined by a systolic blood pressure (SBP) >= 150 mmHg and/or diastolic blood pressure (DBP) >= 100 mmHg with or without antihypertensive medication; NOTE: initiation or adjustment of antihypertensive medication(s) is allowed prior to screening
  * Other clinically significant heart disease or vascular disease
* Currently taking medications that have known or definite risk of prolonging the QT interval or inducing Torsades de pointes (TdP); the medication must be discontinued or switched to a safe alternative medication prior to starting treatment; specific exception is allowed for patients on long-standing medications that have risk of prolonging QT interval or inducing TdP if screening ECG does not indicate a prolonged QT abnormality
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat or dexamethasone (e.g. ulcerative disease uncontrolled nausea, vomiting, malabsorption syndrome, obstruction, or stomach and/or small bowel resection)
* Unresolved diarrhea >= Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or a medical condition associated with chronic diarrhea (such as irritable bowel syndrome, inflammatory bowel disease)
* Major surgery =< 14 days prior to starting study treatment or side effects of surgery that have not recovered to < CTCAE grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cowan, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone: Patients undergo collection of blood and/or bone marrow samples for testing via in vitro chemosensitivity assay. Regardless of assay results, patients receive panobinostat PO on days 1, 3, 5, 15, 17, and 19, and carfilzomib IV and dexamethasone PO on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone
Number analyzed (Participants) | 9
Age, Customized [Median (Full Range); unit: years] | 67 [49 to 72]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6
  Female | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Prior therapy regimes [Median (Full Range); unit: number of regimens] | 5 [2 to 9]
Prior autologous transplant [Number; unit: percentage of participants] | 88.9
Revised ISS Stage [Median (Full Range); unit: ISS Stage] — Revised ISS is the Revised International Staging System, which is used to stage multiple myeloma at diagnosis. It takes into account a patient's albumin, beta-2-microglobulin, lactate dehydrogenase levels, and chromosomal abnormalities detected by FISH to predict survival. There are three stages: I, II, and III. The lower the stage, the longer the progression-free survival.
  ISS Stage | 2.5 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response, by Subject
Description: Assessed using the International Myeloma Working Group Uniform Response Criteria for Multiple Myeloma. Key: 1 = very good partial response (VGPR); 2 = partial response (PR); 3 = minimal response (MR); 4 = stable disease (SD); 5 = progressive disease (PD). Please see IC50 and CI results in the other primary outcome measures.
Time Frame: 14 months
Measure: Number; unit: IMWG Uniform Response Grade
Arm/Group | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone
Number analyzed (Participants) | 9
IMWG Uniform Response Grade
  Subject MM-82 | 4
  Subject MM-91 | 2
  Subject MM-92 | 2
  Subject MM-95 | 1
  Subject MM-96 | 1
  Subject MM-98 | 1
  Subject MM-99 | 3
  Subject MM-109 | 4
  Subject M-111 | 1

2. Primary Outcome: Multiple Myeloma Cells In-vitro Drug Sensitivity to Panobinostat, by Subject
Description: Multiple myeloma cells are added to assay with panobinostat. Cell viability and IC50 is determined. IC50 is the inhibitory concentration that kills 50% of cells. Results are reported in concentrations E-9.
Time Frame: At baseline
Measure: Number; unit: nM
Arm/Group | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone
Number analyzed (Participants) | 9
nM
  Subject MM-82 | 3.8
  Subject MM-91 | 5.9
  Subject MM-92 | 2.6
  Subject MM-95 | 19.8
  Subject MM-96 | 1.3
  Subject MM-98 | 4.4
  Subject MM-99 | 8.5
  Subject MM-109 | 13.6
  Subject MM-111 | 2.0

3. Primary Outcome: Multiple Myeloma Cells In-vitro Drug Sensitivity to Carfilzomib, by Subject
Description: Multiple myeloma cells are added to assay with carfilzomib. Cell viability and IC50 is determined. IC50 is the inhibitory concentration that kills 50% of cells.
Time Frame: At baseline
Measure: Number; unit: nM
Arm/Group | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone
Number analyzed (Participants) | 9
nM
  Subject MM-82 | 17.5
  Subject MM-91 | 0.479
  Subject MM-92 | 0.03
  Subject MM-95 | 0.269
  Subject MM-96 | 0.0048
  Subject MM-98 | 0.159
  Subject MM-99 | 0.159
  Subject MM-109 | 0.108
  Subject MM-111 | 0.0152

4. Primary Outcome: Multiple Myeloma Cells In-vitro Drug Sensitivity to Dexamethasone, by Subject
Description: Multiple myeloma cells are added to assay with dexamethasone. Cell viability and IC50 is determined. IC50 is the inhibitory concentration that kills 50% of cells. Results are reported in concentrations E-6.
Time Frame: At baseline
Population: Results for subject MM-92 were not reported.
Measure: Number; unit: uM
Arm/Group | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone
Number analyzed (Participants) | 8
uM
  Subject MM-82 | 3.7
  Subject MM-91 | 10.9
  Subject MM-95 | 7
  Subject MM-96 | 1.1
  Subject MM-98 | 14.8
  Subject MM-99 | 8.6
  Subject MM-109 | 80
  Subject MM-111 | 1.1

5. Primary Outcome: Synergy of Panobinostat and Carfilzomib in Combination, Per Subject.
Description: Concentration of carfilzomib and panobinostat in combination leading to 90% growth inhibition of multiple myeloma cells in-vitro. The combination index (CI) is calculated using formula: CI = ([D1] in the combination / [D1] alone) + ([D2] in the combination / [D2] alone). Key: CI = 1 no synergy; CI<1 synergy; CI>1 antagonism.
Time Frame: At baseline
Population: CI score was not reported for subject MM-82.
Measure: Number; unit: Combination index
Arm/Group | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone
Number analyzed (Participants) | 8
Combination index
  Subject MM-91 | 2.5
  Subject MM-92 | 2.4
  Subject MM-95 | 0.3
  Subject MM-96 | 2.2
  Subject MM-98 | 2.6
  Subject MM-99 | 1.8
  Subject MM-109 | 1.7
  Subject MM-111 | 62.2

6. Primary Outcome: Synergy of Panobinostat and Dexamethasone in Combination, Per Subject
Description: Concentration of panobinostat and dexamethasone in combination leading to 90% growth inhibition of multiple myeloma cells in-vitro. The combination index (CI) is calculated using formula: CI = ([D1] in the combination / [D1] alone) + ([D2] in the combination / [D2] alone). Key: CI = 1 no synergy; CI<1 synergy; CI>1 antagonism.
Time Frame: At baseline
Population: CI score was not reported for subject MM-82
Measure: Number; unit: CI score
Arm/Group | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone
Number analyzed (Participants) | 8
CI score
  Subject MM-91 | 1.3
  Subject MM-92 | 2.6
  Subject MM-95 | 1.4
  Subject MM-96 | 0.6
  Subject MM-98 | 1.2
  Subject MM-99 | 0.9
  Subject MM-109 | 4.6
  Subject MM-111 | 1.2

ADVERSE EVENTS:
Time Frame: Adverse events after any administration of the study drug through 30 days after the last administration of therapy will be recorded and followed until resolution.
Description: Only non-hematologic toxicities ≥ grade 3 will be reported as adverse events. Hospitalizations or prolongation of hospitalizations for protocol-schedule procedures, blood product transfusions, or social reasons (i.e. awaiting transport home) will not be considered a SAE.
Arm/Group | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone (N=9)
Non-ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
Fracture, pathologic (Injury, poisoning and procedural complications) | 1 (1)
Fracture, non-pathologic (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemo Assay and Treatment With Panobinostat, Carfilzomib, and Dexamethasone (N=9)
Hypertension (Vascular disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was limited by lower accrual than expected due to: competing studies, other investigators' treatment preferences, and ultimately, the departure of the initial PI from the institution. Because of PI's departure and lab closure, the study closed to accrual after the 9th patient enrolled. Because only 9 subjects were enrolled and some in-vitro assay results are unavailable, it is difficult to analyze the in-vitro assay results and determine the parameters that predict disease response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT03256045/Prot_SAP_001.pdf